CLINICAL TRIAL: NCT00744497
Title: A Randomized Double-Blind Phase 3 Trial Comparing Docetaxel Combined With Dasatinib to Docetaxel Combined With Placebo in Castration-Resistant Prostate Cancer
Brief Title: Randomized Study Comparing Docetaxel Plus Dasatinib to Docetaxel Plus Placebo in Castration-resistant Prostate Cancer
Acronym: READY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CA180-227; 2008-000701-11 (EudraCT Number)
Record Dates: First submitted 2008-08-29; First posted 2008-09-01 (Estimated); Results first posted 2014-02-06 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-08

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Dasatinib; Docetaxel; Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Participants received placebo, given orally once daily, plus docetaxel, 75 mg/m^2, given intravenously every 3 weeks as a 1-hour infusion, plus prednisone, 5 mg, given orally twice daily
  Interventions: Drug: Placebo; Drug: Docetaxel; Drug: Prednisone
- Dasatinib (Active Comparator): Participants received dasatinib, 100 mg, orally once daily plus docetaxel, 75 mg/m^2, given intravenously every 3 weeks as a 1-hour infusion, plus prednisone, 5 mg, given orally twice daily
  Interventions: Drug: Dasatinib; Drug: Docetaxel; Drug: Prednisone

INTERVENTIONS:
Drug: Placebo
  Arms: Placebo
Drug: Dasatinib
  Other Names: Sprycel; BMS-354825
  Arms: Dasatinib
Drug: Docetaxel
Drug: Prednisone

SUMMARY:
The purpose of this study is to determine whether survival can be prolonged in patients with castration-resistant prostate cancer who receive dasatinib with docetaxel and prednisone.

ELIGIBILITY:
Inclusion Criteria:

* History of histologically diagnosed prostate cancer
* Evidence of metastatic disease by any 1 of the following: computed tomography scan, magnetic resonance imaging, bone scan, or skeletal survey
* Evidence of progression, as defined by 1 of the following: rising prostate specific antigen levels at least 1 week apart with the final value being >=2 ng/mL; progression of measurable nodal or visceral disease, with nodal lesions >=20 mm and visceral lesions measurable per response evaluation criteria for solid tumors (Response Evaluation in Solid Tumors, version 1); 2 or more lesions appearing on bone scan compared with previous scan; or local recurrence in the prostate or prostate bed
* Maintaining castrate status: Participants who have not undergone surgical orchiectomy should have received and continue on medical therapies, such as gonadotropin releasing hormone analogs, to maintain castrate levels of serum testosterone <=50 ng/dL
* Eastern Cooperative Oncology Group Performance Status of 0 to 2
* At least 4 weeks since an investigational agent prior to starting study therapy
* At least 8 weeks since radioisotope therapy prior to starting study therapy
* Recovery from any local therapy including surgery or radiation/radiotherapy for a minimum of 7 days prior to starting study therapy
* Required initial laboratory values: white blood cell count >=3,000/mm^3; absolute neutrophil count >=1,500/mm^3; platelet count >=100,000/mm^3; creatinine level <=1.5*upper limit of normal (ULN); bilirubin <=ULN; aspartate aminotransferase <=2.5*ULN; alanine aminotransferase <=2.5*ULN.

Exclusion Criteria:

* Symptomatic brain metastases or leptomeningeal metastases
* Clinically significant cardiovascular disease, including myocardial infarction; ventricular tachyarrhythmia within 6 months; prolonged QTc >450 msec; ejection fraction <40%; or major conduction abnormality, unless a cardiac pacemaker is present
* Pleural or pericardial effusion of any Common Terminology Criteria (CTC) grade
* Peripheral neuropathy CTC Grade >=2
* Currently active second malignancy other than nonmelanoma skin cancers. Participants are not considered to have a currently active malignancy if they have completed therapy and are now considered (by their physician) to be at less than 30% risk for relapse
* Uncontrolled intercurrent illness including ongoing or active infection, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* HIV infection-positive patients receiving combination antiretroviral therapy
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to the investigational agents
* Receipt of any other investigational agents for the treatment of prostate cancer
* Prior cytotoxic chemotherapy in the metastatic setting, with the exception of estramustine
* Patients may continue on a daily multivitamin but must discontinue all other herbal, alternative, and food supplements before enrollment
* Ketoconazole must be discontinued 4 weeks prior to starting study therapy
* Antiandrogens must be discontinued prior to starting study therapy. Patients with a history of response to an antiandrogen and subsequent progression while on that antiandrogen should be assessed for antiandrogen withdrawal response for 4 weeks. Observation for antiandrogen withdrawal response is not necessary for those who have never responded to antiandrogens
* Bisphosphonates must not be initiated within 28 days prior to starting study therapy
* QT prolonging agents strongly associated with torsade de pointes.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1930 (Actual)
Dates: Start 2008-10; Primary Completion 2012-08 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (160):
- United States (42):
  - University Of South Alabama / Mitchell Cancer Institute, Mobile, Alabama
  - Southern Cancer Center, Mobile, Alabama
  - Alaska Clinical Research Center, Llc, Anchorage, Alaska
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Compassionate Cancer Care Medical Group, Inc., Corona, California
  - Desert Hematology Oncology Medical Group, Rancho Mirage, California
  - Compassionate Cancer Care Medical Group Inc, Riverside, California
  - Sharp Clinical Oncology Research, San Diego, California
  - Va San Diego Healthcare System, San Diego, California
  - Edward Alexson, Md, Inc., Santa Ana, California
  - Connecticut Oncology Group, Middletown, Connecticut
  - Va Connecticut Healthcare System, West Haven, Connecticut
  - Gwinnett Hospital System Inc., Lawrenceville, Georgia
  - University Of Chicago, Chicago, Illinois
  - Midwestern Regional Medical Center, Zion, Illinois
  - Fort Wayne Medical Oncology And Hematology Inc, Fort Wayne, Indiana
  - Cancer Center Of Kansas, Wichita, Kansas
  - Maine Center For Cancer Medicine, Scarborough, Maine
  - Tufts Medical Center, Boston, Massachusetts
  - Jackson Oncology Associates, Pllc, Jackson, Mississippi
  - North Mississippi Hematology And Oncology Associates, Ltd, Tupelo, Mississippi
  - New York Oncology Hematology, Pc, Albany, New York
  - Samuel S. Stratton Vamc, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Piedmont Hematology Oncology Associates, Pllc, Winston-Salem, North Carolina
  - Summa Health System, Akron, Ohio
  - Mid Ohio Oncology/Hematology, Inc,Dba, Columbus, Ohio
  - Providence Portland Med Ctr, Portland, Oregon
  - Regional Hemetology Oncology, Pc, Langhorne, Pennsylvania
  - Upmc Cancer Pavilion, Pittsburgh, Pennsylvania
  - Va Pittsburgh Healthcare System, Pittsburgh, Pennsylvania
  - Associates In Hematology & Oncology, P.C., Upland, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island
  - Cancer Centers Of The Carolinas, Greenville, South Carolina
  - Boston Baskin Cancer Foundation, Memphis, Tennessee
  - Cancer Specialists Of South Texas, Pa, Corpus Christi, Texas
  - The University Of Texas Md Anderson Cancer Center, Houston, Texas
  - Providence Regional Cancer System, Lacey, Washington
  - University Of Washington, Seattle, Washington
  - Dean Hematology And Oncology Clinic, Madison, Wisconsin
- Argentina (9):
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Caba, Buenos Aires
  - Local Institution, Capital Federal, Buenos Aires
  - Local Institution, La Plata, Buenos Aires
  - Local Institution, Ramos Mejía, Buenos Aires
  - Local Institution, Cipolletti, Río Negro Province
  - Local Institution, Rosario, Santa Fe Province
  - Local Institution, San Miguel de Tucumán, Tucumán Province
  - Local Institution, Cordaba
- Australia (11):
  - Local Institution, Coffs Harbour, New South Wales
  - Local Institution, Lismore, New South Wales
  - Local Institution, Port Macquarie, New South Wales
  - Local Institution, Sydney, New South Wales
  - Local Institution, Douglas, Queensland
  - Local Institution, Milton, Queensland
  - Local Institution, Kurralta Park, South Australia
  - Local Institution, Hobart, Tasmania
  - Local Institution, Frankston, Victoria
  - Local Institution, Ringwood, Victoria
  - Local Institution, Fremantle, Western Australia
- Brazil (7):
  - Local Institution, Salvador, Estado de Bahia
  - Local Institution, Rio de Janeiro, Rio de Janeiro
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, Barretos, São Paulo
  - Local Institution, Campinas, São Paulo
  - Local Institution, Jaú, São Paulo
  - Local Institution, Santo André, São Paulo
- Canada (13):
  - Local Institution, Edmonton, Alberta
  - Local Institution, Abbottsford, British Columbia
  - Local Institution, Moncton, New Brunswick
  - Local Institution, Greater Sudbury, Ontario
  - Local Institution, Ottawa, Ontario
  - Local Institution, Owen Sound, Ontario
  - Local Institution, Thunder Bay, Ontario
  - Local Institution, Greenfield Park, Quebec
  - Local Institution, Montreal, Quebec
  - Local Institution, Rimouski, Quebec
  - Local Institution, Sherbrooke, Quebec
  - Local Institution, Regina, Saskatchewan
  - Local Institution, Saskatoon, Saskatchewan
- Czechia (3):
  - Local Institution, Brno
  - Local Institution, Hradec Králové
  - Local Institution, Prague
- Finland (2):
  - Local Institution, Turku
  - Local Institution, Vaasa
- France (7):
  - Local Institution, Avignon
  - Local Institution, Besançon
  - Local Institution, Caen
  - Local Institution, Créteil
  - Local Institution, Paris
  - Local Institution, Saint-Genis-Laval
  - Local Institution, Strasbourg
- Germany (6):
  - Local Institution, Aachen
  - Local Institution, Berlin
  - Local Institution, Erlangen
  - Local Institution, Essen
  - Local Institution, Kirchheim
  - Local Institution, Markkleeberg
- Local Institution, Athens, Greece
- Hungary (3):
  - Local Institution, Budapest
  - Local Institution, Kecskemét
  - Local Institution, Zalaegerszeg
- India (6):
  - Local Institution, Trivandrum, Kerala
  - Local Institution, Mumbai, Maharashtra
  - Local Institution, Pune, Maharashtra
  - Local Institution, Ahmedabad
  - Local Institution, Jaipur
  - Local Institution, Kolkata
- Ireland (3):
  - Local Institution, Cork, Cork
  - Local Institution, Dublin, Dublin
  - Local Institution, Tallaght, Dublin
- Italy (7):
  - Local Institution, Arezzo
  - Local Institution, Genova
  - Local Institution, Lecce
  - Local Institution, Milan
  - Local Institution, Napoli
  - Local Institution, Perugia
  - Local Institution, Roma
- Mexico (10):
  - Local Institution, Tijuana, Estado de Baja California
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Zapopan, Jalisco
  - Local Institution, Df, Mexico City
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Tlalpan, Mexico City
  - Local Institution, Monterrey, Nuevo León
  - Local Institution, México, Querétaro
  - Local Institution, Huixquilucan, State of Mexico
  - Local Institution, Toluca, State of Mexico
- Local Institution, Stavanger, Norway
- Peru (2):
  - Local Institution, Lima, Lima Province
  - Local Institution, Callao, Provincia Constitucional del Callao
- Poland (3):
  - Local Institution, Bialystok
  - Local Institution, Lodz
  - Local Institution, Warsaw
- Romania (3):
  - Local Institution, Baia Mare
  - Local Institution, Cluj-Napoca
  - Local Institution, Timisoara, Timis
- Russia (2):
  - Local Institution, Moscow
  - Local Institution, Saint Petersburg
- South Africa (3):
  - Local Institution, Bloemfontein, Free State
  - Local Institution, Pretoria, Gauteng
  - Local Institution, Saxonwold, Gauteng
- Local Institution, Seoul, South Korea
- Spain (6):
  - Local Institution, Barcelona
  - Local Institution, Gijón
  - Local Institution, Madrid
  - Local Institution, Santander
  - Local Institution, Seville
  - Local Institution, Valencia
- Sweden (4):
  - Local Institution, Kungälv
  - Local Institution, Sundsvall
  - Local Institution, Uppsala
  - Local Institution, Vaxjo
- United Kingdom (5):
  - Local Institution, Essex, Essex
  - Local Institution, Cardiff, Glamorgan
  - Local Institution, London, Middlesex
  - Local Institution, Sutton, Surrey
  - Local Institution, Leeds, West Yorkshire

REFERENCES:
- [Derived] de Liano AG, Reig O, Mellado B, Martin C, Rull EU, Maroto JP. Prognostic and predictive value of plasma testosterone levels in patients receiving first-line chemotherapy for metastatic castrate-resistant prostate cancer. Br J Cancer. 2014 Apr 29;110(9):2201-8. doi: 10.1038/bjc.2014.189. Epub 2014 Apr 10. PMID 24722180
- [Derived] Araujo JC, Trudel GC, Saad F, Armstrong AJ, Yu EY, Bellmunt J, Wilding G, McCaffrey J, Serrano SV, Matveev VB, Efstathiou E, Oudard S, Morris MJ, Sizer B, Goebell PJ, Heidenreich A, de Bono JS, Begbie S, Hong JH, Richardet E, Gallardo E, Paliwal P, Durham S, Cheng S, Logothetis CJ. Docetaxel and dasatinib or placebo in men with metastatic castration-resistant prostate cancer (READY): a randomised, double-blind phase 3 trial. Lancet Oncol. 2013 Dec;14(13):1307-16. doi: 10.1016/S1470-2045(13)70479-0. Epub 2013 Nov 8. PMID 24211163
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1930 participants enrolled, 1522 randomized to a treatment group (762 dasatinib, 760 placebo). 408 not randomized. Reasons for non-randomization include 7 adverse events, 42 withdrew consent, 6 deaths, 2 lost to follow up, 3 poor/non compliance, 332 no longer met study criteria, 1 administrative reason by sponsor, and 15 non-specified reasons.
Period: Overall Study
Arm/Group | Placebo | Dasatinib
Started | 760 (Randomized) | 762 (Randomized)
Received Treatment | 757 | 761
Completed | 0 | 0
Not Completed | 760 | 762
Not completed — Withdrawal by Subject | 21 | 18
Not completed — Death | 11 | 9
Not completed — Lost to Follow-up | 4 | 2
Not completed — Poor compliance/noncompliance | 9 | 5
Not completed — No longer meets study criteria | 7 | 3
Not completed — Administrative Reason By Sponsor | 25 | 8
Not completed — Disease progression | 312 | 219
Not completed — Study drug toxicity | 68 | 141
Not completed — Adverse event unrelated to study drug | 78 | 122
Not completed — Patient requested to stop study drug | 65 | 80
Not completed — Maximum clinical benefit | 141 | 142
Not completed — Not defined | 19 | 13

BASELINE CHARACTERISTICS:
Population: All participants who were randomized to receive any treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dasatinib | Total
Number analyzed (Participants) | 760 | 762 | 1522
Age, Customized [Number; unit: participants]
  Younger than 65 years | 263 | 251 | 514
  65 to younger than 75 years | 323 | 333 | 656
  75 years or older | 174 | 178 | 352
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 760 | 762 | 1522
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 56 | 55 | 111
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 34 | 23 | 57
  White | 645 | 656 | 1301
  Other | 24 | 27 | 51
Type of metastatic disease [Number; unit: Participants]
  Bone disease only | 286 | 307 | 593
  Visceral/nodal disease only | 73 | 80 | 153
  Both bone and visceral/nodal disease | 399 | 373 | 772
  No evidence of metastatic disease | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival: Time From Randomization to Date of Death
Description: Overall survival is defined as time in months from the randomization date to the date of death due to any cause (in the randomized population). If the patient did not die, survival was censored on the last date he or she was known to be alive.
Time Frame: From randomization to death or date of last contact (maximum reached: 45 months)
Population: All participants who were randomized to receive any treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo | Dasatinib
Number analyzed (Participants) | 760 | 762
Months | 21.2 [20.0 to 23.4] | 21.5 [20.3 to 22.8]
Statistical Analysis 1: Comparison: Placebo vs Dasatinib; Confidence intervals for median overall survival calculated using Brookmeyer and Crowley method. Compared survival in arms by 2-sided, alpha=0.0447 level, log-rank test, stratified by bisphosphonate intake (yes/no) and urinary N-telopeptide category (<60 vs ≥60 nmol/mmol creatinine) defined at randomization. Null hypothesis was survival equal in both arms. Power calculations were that ≥858 deaths would lead to ≥90% power at 5% level for rejecting null hypothesis, given true hazard ratio of 0.8; Test type: Superiority or Other; p = 0.9009, Log Rank — An interim analysis on survival was performed and the final test was corrected for multiplicity; Hazard Ratio (HR) = 0.99, 95.53% CI 2-sided [0.87 to 1.13]

2. Secondary Outcome: Percentage of Participants With an Objective Tumor Response by Modified Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Objective tumor response rate=the percentage of randomized participants with a best tumor response of partial (PR) or complete response (CR), within 42 days of end of dosing, divided by total number of patients who were evaluable (with at least 1 target lesion at baseline). By RECIST: CR=disappearance of clinical and radiologic evidence of target and nontarget lesions confirmed by another evaluation at least 6 weeks later. PR=a >30% or greater decrease in the sum of longest diameter (LD) of target lesions in reference to the baseline sum LD confirmed by another evaluation at least 6 weeks later. Stable disease=neither sufficient increase to qualify for PD nor shrinkage to qualify for PR, and at least 8 weeks since start of study therapy. Progressive disease=a 20% or greater increase in sum of LD of all target lesions, taking as reference the smallest sum of LD at or following baseline, or unequivocal progression on existing nontarget lesions, or new lesions are present.
Time Frame: At baseline and every 12 weeks thereafter to end of treatment, at end of treatment, and at follow-up (within 42 days of end of dosing)
Population: Participants with at least 1 target lesion at baseline
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Dasatinib
Number analyzed (Participants) | 383 | 381
Percentage of participants | 31.85 [27.21 to 36.78] | 30.45 [25.86 to 35.34]
Statistical Analysis 1: Comparison: Placebo vs Dasatinib; Since superiority of the dasatinib treatment group was not demonstrated for Overall Survival, secondary endpoints were not tested. The odds ratio is presented for experimental to control group; Test type: Superiority or Other; Odds Ratio (OR) = 0.935, 95% CI 2-sided [0.688 to 1.271]

3. Secondary Outcome: Time to First Skeletal-related Event (SRE)
Description: Time to first SRE is defined as the time in months from the date of randomization to the date of first SRE (unless SRE occurred while the patient was undergoing subsequent cancer therapy). Participants with a first SRE while on subsequent cancer therapy, those who died without a reported SRE, and those who did not have an SRE were censored on the date of their last SRE assessment prior to start of subsequent cancer therapy, if any. Participants who had no SRE assessments were censored on the day they were randomized.
Time Frame: From day of randomization to date of first SRE or to last SRE assessment, if subsequent cancer therapy begun or no SRE (maximum reached: 42 months)
Population: All participants who were randomized to receive any treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo | Dasatinib
Number analyzed (Participants) | 760 | 762
Months | 31.1 [28.8 to NA] — NA=Not estimable; insufficient number of participants with events | NA [NA to NA] — NA=Not estimable; insufficient number of participants with events
Statistical Analysis 1: Comparison: Placebo vs Dasatinib; Since superiority of the dasatinib treatment group was not demonstrated for Overall Survival, secondary endpoints were not tested. The hazard ratio is presented for experimental to control group; Test type: Superiority or Other; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.64 to 1.02]

4. Secondary Outcome: Percentage of Participants With A Reduction in Urinary N-telopeptide (uNTx) Level From Baseline
Description: The percentage of participants who had an on-study uNTx value confirmed (at least 3 weeks later) within normal limits (or ≥3 and <60 nmol/mmol creatinine, if normal limits were missing) or an on-study uNTx level reduction from baseline of ≥35%, even when on-study uNTx value remained abnormal.
Time Frame: At baseline, prior to each docetaxel infusion (every 3 weeks) to end of treatment, at end of treatment, and at follow-up (within 14 days of end of dosing)
Population: Participants who entered the study with baseline urinary N-telopeptide values higher than the upper limit of normal (ULN), or ≥60 nmol/mmol creatinine, if ULN was missing
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Dasatinib
Number analyzed (Participants) | 335 | 321
Percentage of participants | 60.60 [55.14 to 65.86] | 66.04 [60.58 to 71.21]
Statistical Analysis 1: Comparison: Placebo vs Dasatinib; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Odds Ratio (OR) = 1.280, 95% CI 2-sided [0.930 to 1.763]

5. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the time from the randomization date until the date of earliest evidence of disease progression or death, for participants who progressed or died before subsequent cancer therapy. Those who progressed or died while on subsequent cancer therapy and those who did not die or progress were censored at their last radiologic bone scan/imaging, skeletal related-event, or tumor assessment or at measurement of prostate specific antigen levels, whichever occurred last prior to start of subsequent cancer therapy ,if any. Participants with no assessments were censored on the day of randomization.
Time Frame: From day of randomization to disease progression or death (or to last clinical assessment, if subsequent cancer therapy started or no progression or death) (maximum reached: approximately 43 months)
Population: All participants who were randomized to receive any treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo | Dasatinib
Number analyzed (Participants) | 760 | 762
Months | 11.1 [10.8 to 11.7] | 11.8 [11.1 to 13.4]
Statistical Analysis 1: Comparison: Placebo vs Dasatinib; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.82 to 1.05]

6. Secondary Outcome: Time to Prostate Specific Antigen (PSA) Progression
Description: PSA progression is defined as the time from randomization to the date of the first PSA level measurement that led to confirmed PSA progression, for participants who had not started subsequent cancer therapy. For participants who did not progress or who progressed on cancer therapy, PSA progression is defined as the time from randomization to the date of the last PSA level measurement before the start of cancer therapy, if any. Participants who had no on-study PSA level measurements were censored on the day they were randomized.
Time Frame: From randomization to date of first PSA measurement leading to confirmed PSA progression (or to last bone scan assessment, if no progression or if cancer therapy started) (maximum reached: 30 months)
Population: All participants who were randomized to receive any treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo | Dasatinib
Number analyzed (Participants) | 760 | 762
Months | 6.9 [6.5 to 7.4] | 7.2 [6.6 to 7.9]
Statistical Analysis 1: Comparison: Placebo vs Dasatinib; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.79 to 1.01]

7. Secondary Outcome: Percentage of Participants With a Reduction in Pain Intensity From Baseline
Description: The percentage of participants with a reduction in pain intensity from baseline was defined as the number of participants who achieved a 30% or more decrease in pain intensity from baseline for at least 2 consecutive pain assessments (at least 14 days apart) within 14 days of end of dosing divided by the number of randomized participants who had a baseline pain intensity of at least 2. Pain intensity was assessed based on question 3 of the brief pain inventory questionnaire.
Time Frame: At baseline, prior to each docetaxel infusion (every 3 weeks), at end of treatment, and at follow-up (within 14 days of end of dosing)
Population: Participants with a baseline pain intensity of 2 or greater
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Dasatinib
Number analyzed (Participants) | 467 | 419
Percentage of participants | 71.52 [67.19 to 75.57] | 66.59 [61.85 to 71.09]
Statistical Analysis 1: Comparison: Placebo vs Dasatinib; Since superiority of the dasatinib treatment group was not demonstrated for Overall Survival, secondary endpoints were not tested. The odds ratio is presented for of experimental to control group; Test type: Superiority or Other; Odds Ratio (OR) = 0.791, 95% CI 2-sided [0.594 to 1.052]

8. Other Pre Specified Outcome: Number of Participants With Serious Adverse Event (SAEs), Drug-related SAEs, Drug-related AEs, Drug-related AEs Leading to Discontinuation, and All Deaths
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Drug-related=having certain, probable, possible, or missing relationship to study drug
Time Frame: Continuously throughout study to <=30 days after last dose of study drug; included AEs with an onset date >= day 1 and <= last dose date + 30 days
Population: All participants who received treatment
Measure: Number; unit: Participants
Arm/Group | Placebo | Dasatinib
Number analyzed (Participants) | 757 | 761
Participants
  All deaths | 505 | 506
  Deaths within 30 days of end of treatment | 50 | 79
  All SAEs | 317 | 381
  Drug-related SAEs | 90 | 150
  All Drug-related AEs | 482 | 553
  Drug-related AEs leading to discontinuation | 76 | 144

9. Other Pre Specified Outcome: Number of Participants With Drug-Related Adverse Events (AEs) of Special Interest
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. AEs of Special Interest=recognized events in other agents within this drug class or events for which safety data from nonclinical and clinical studies with dasatinib indicate that careful evaluation is warranted. Drug-related=having certain, probable, possible, or missing relationship to study drug. Drug-related AEs of Special Interest are identified by the medical and safety representatives of the sponsor based on MedDRA preferred terms or laboratory data. ANC=absolute neutrophil count.
Time Frame: as for outcome 8
Population: All participants who received treatment
Measure: Number; unit: Participants
Arm/Group | Placebo | Dasatinib
Number analyzed (Participants) | 757 | 761
Participants
  Diarrhea | 167 | 229
  Nausea/vomiting | 127 | 170
  Fatigue | 216 | 236
  Myalgias/arthralgias | 29 | 29
  Rash | 46 | 72
  Gastrointestinal tract bleeding | 6 | 14
  Central nervous system bleeding | 1 | 2
  Other hemorrhage | 14 | 24
  Pulmonary arterial hypertension | 0 | 0
  Fluid retention: Superficial edema | 77 | 76
  Fluid retention: Pleural effusion | 13 | 87
  Fluid retention: Other | 37 | 52

10. Other Pre Specified Outcome: Number of Participants With Abnormalities in Results of Clinical Laboratory Tests in Hematology
Description: Abnormalities were graded according to the Common Toxicity Criteria (CTC), version 3.0, of the National Cancer Institute. CTC are graded from 1 (least severe) to 4 (life threatening ). Grade 3 and 4 criteria are defined as follows: Absolute neutrophil count, Grade 3, neutrophils <1.0-0.5*10^9/L; Grade 4, <0.5*10^9/L. Hemoglobin, Grade 3, <4.9-4.0 mmol/L; Grade 4, <4.0 mmol/L. Platelets, Grade 3, <50.0-25.0*10^9/L; Grade 4, <25.0*10^9/L. Leukocytes, Grade 3, <2.0-1.0*10^9/L; Grade 4, <1.0*10^9/L.
Time Frame: At baseline, within 3 days prior to each infusion of docetaxel (each cycle) and at end of treatment. If docetaxel is discontinued, every other cycle.
Population: All participants who received treatment
Measure: Number; unit: Participants
Arm/Group | Placebo | Dasatinib
Number analyzed (Participants) | 757 | 761
Participants
  Absolute neutrophil count (All grades) | 84 | 161
  Absolute neutrophil count (Grades 3 and 4) | 41 | 46
  Hemoglobin (All grades) | 712 | 720
  Hemoglobin (Grades 3 and 4) | 44 | 59
  Platelets (All grades) | 108 | 100
  Platelets (Grades 3 and 4) | 6 | 3
  Leukocytes (All grades) | 128 | 149
  Leukocytes (Grades 3 and 4) | 32 | 30

11. Other Pre Specified Outcome: Number of Participants With Abnormalities in Results of Clinical Laboratory Tests Assessing Liver Function, Renal Function, and Electrolytes
Description: ALP=alkaline phosphatase; ALT=alanine aminotransferase; AST=aspartate aminotransferase; ULN=upper limit of normal. Abnormalities were graded according to the Common Toxicity Criteria (CTC), version 3.0, of the National Cancer Institute. CTC are graded from 1 (least severe) to 4 (life threatening). ALP, ALT, and AST, Grade 3, >5.0-20.0*ULN; Grade 4, >20.0*ULN. Total bilirubin, Grade 3, >3.0-10.0*ULN; Grade 4, >10.0*ULN. Creatinine, Grade 3, >3.0-6.0*ULN; Grade 4, >6.0*ULN. Hypercalcemia(serum calcium, mmol/L), Grade 3, >3.1-3.4; Grade 4, >3.4. Hypocalcemia (serum calcium, mmol/L), Grade 3, <1.75-1.5; Grade 4, <1.5. Hyperkalemia(serum calcium, mmol/L), Grade 3, >6.0-7.0; Grade 4, >7.0. Hypokalemia(serum calcium, mmol/L), Grade 3, <3.0-2.5; Grade 4, <2.5. Hypernatremia (serum calcium, mmol/L), Grade 3, >155-160; Grade 4, >160. Hyponatremia (serum sodium, mmol/L), Grade 3, <130-120; Grade 4, <120. Phosphorus (serum sodium, mmol/L), Grade 3, <0.6-0.3; Grade 4, <0.3.
Time Frame: At baseline, within 3 days prior to each infusion of docetaxel (each cycle), to end of treatment. If docetaxel is discontinued, every other cycle.
Population: All participants who received treatment
Measure: Number; unit: Participants
Arm/Group | Placebo | Dasatinib
Number analyzed (Participants) | 757 | 761
Participants
  ALP (All grades) | 447 | 375
  ALP (Grades 3 and 4) | 91 | 68
  ALT (All grades) | 186 | 256
  ALT (Grades 3 and 4) | 5 | 6
  AST (All grades) | 212 | 266
  AST (Grades 3 and 4) | 4 | 5
  Total bilirubin (All grades) | 49 | 41
  Total bilirubin (Grades 3 and 4) | 1 | 3
  Creatinine (All grades) | 153 | 184
  Creatinine (Grades 3 and 4) | 3 | 5
  Hypercalcemia (All grades) | 56 | 34
  Hypercalcemia (Grades 3 and 4) | 1 | 1
  Hypocalcemia (All grades) | 308 | 377
  Hypocalcemia (Grades 3 and 4) | 23 | 25
  Hyperkalemia (All grades) | 164 | 152
  Hyperkalemia (Grades 3 and 4) | 11 | 14
  Hypokalemia (All grades) | 107 | 152
  Hypokalemia (Grades 3 and 4) | 6 | 16
  Hypernatremia (All grades) | 93 | 101
  Hypernatremia (Grades 3 and 4) | 0 | 0
  Hyponatremia (All grades) | 230 | 241
  Hyponatremia (Grades 3 and 4) | 36 | 43
  Phosporus (All grades) | 189 | 257
  Phosphorus (Grades 3 and 4) | 43 | 93

12. Other Pre Specified Outcome: Number of Participants With Abnormal Results in Urinalysis
Description: Abnormal=positive, defined as the presence of >=30 mg/dL of protein; a small, moderate, or large amount of blood; or >0 g/dL glucose in urine. BL=baseline; neg=negative
Time Frame: as for outcome 11
Population: All participants who received treatment.
Measure: Number; unit: Participants
Arm/Group | Placebo | Dasatinib
Number analyzed (Participants) | 757 | 761
Participants
  Protein, urine: postive | 246 | 336
  Blood, urine: positive | 289 | 307
  Glucose, urine: positive | 179 | 154

13. Other Pre Specified Outcome: Number of Participants by Maximal On-study Fridericia-corrected QTc Interval
Description: QTc interval measured by electrocardiogram (ECG). Although a participant may have had several ECGs, only the longest QTc interval was included.
Time Frame: At baseline, approximately 12 weeks after starting treatment, and then whenever clinically indicated up to within 30 days of end of dosing
Population: All participants who received treatment. n=number evaluable
Measure: Number; unit: Participants
Arm/Group | Placebo | Dasatinib
Number analyzed (Participants) | 757 | 761
Participants
  <450 msecs (n=600, 548) | 550 | 497
  450-500 msecs (n=600, 548) | 43 | 48
  >500 msecs (n=600, 548) | 7 | 3

14. Other Pre Specified Outcome: Number of Participants With Changes From Baseline in Fridericia-corrected QTc Interval
Description: as for outcome 13
Time Frame: as for outcome 13
Population: All participants who received treatment. n=number evaluable
Measure: Number; unit: Participants
Arm/Group | Placebo | Dasatinib
Number analyzed (Participants) | 757 | 761
Participants
  0 to 30 msecs increase (n=591, 540) | 203 | 199
  >30 to 60 msecs increase (n=591, 540) | 52 | 47
  >60 msecs increase (n=591, 540) | 32 | 26
  Decrease (n=591, 540) | 304 | 268

15. Other Pre Specified Outcome: Number of Participants With and Without Pericardial Effusion at Baseline and On-study and With Left Ventricular Ejection Fraction (LVEF) <40% and >=40% On-study
Description: BL=baseline; OS=on-study
Time Frame: At baseline, approximately 12 weeks after start of treatment, and thereafter whenever clinically indicated
Population: All participants who were randomized to receive any treatment
Measure: Number; unit: Participants
Arm/Group | Placebo | Dasatinib
Number analyzed (Participants) | 760 | 762
Participants
  Pericardial effusion at BL/absent OS | 3 | 1
  Pericardial effusion at BL/present OS | 0 | 1
  Pericardial effusion at BL/not reported OS | 1 | 0
  Pericardial effusion absent at BL/ absent OS | 584 | 545
  Pericardial effusion absent at BL/present OS | 24 | 26
  Pericardial effusion absent at BL/not reported OS | 132 | 184
  Pericardial not reported at BL | 16 | 5
  LVEF OS <40% | 2 | 2
  LVEF OS >=40% | 607 | 566
  LVEF not reported OS | 151 | 194

ADVERSE EVENTS:
Time Frame: Day 1 up to 30 days post last dose of study therapy
Description: Study initiated: October 2008; Study Completion: July 2015
Arm/Group | Placebo | Dasatinib
Serious Adverse Events (participants affected / at risk) | 317/757 | 381/761
Other Adverse Events (participants affected / at risk) | 701/757 | 716/761
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=757) | Dasatinib (N=761)
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 4 | 8
Adenosquamous cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 2
Deep vein thrombosis (Vascular disorders) | 10 | 1
Device occlusion (General disorders) | 2 | 0
Diverticulitis (Infections and infestations) | 3 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 21
Empyema (Infections and infestations) | 1 | 0
Enterovesical fistula (Gastrointestinal disorders) | 1 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 1 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 3 | 3
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 1 | 0
Haemoglobinuria (Renal and urinary disorders) | 1 | 0
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 2
Hip fracture (Injury, poisoning and procedural complications) | 1 | 2
Hydronephrosis (Renal and urinary disorders) | 3 | 6
Hypersensitivity (Immune system disorders) | 1 | 3
Hyperthermia (General disorders) | 0 | 1
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 | 0
Hypotension (Vascular disorders) | 8 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 7 | 9
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Nerve root compression (Nervous system disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain (General disorders) | 9 | 7
Paraparesis (Nervous system disorders) | 1 | 0
Peripheral swelling (General disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pyrexia (General disorders) | 14 | 29
Radiation proctitis (Injury, poisoning and procedural complications) | 0 | 4
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Reflux gastritis (Gastrointestinal disorders) | 1 | 0
Renal disorder (Renal and urinary disorders) | 0 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Scrotal abscess (Infections and infestations) | 1 | 0
Shock haemorrhagic (Vascular disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 2
Supraventricular tachycardia (Cardiac disorders) | 2 | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 0
Venous injury (Injury, poisoning and procedural complications) | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 1
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 15 | 21
Astrocytoma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder neck obstruction (Renal and urinary disorders) | 0 | 1
Bladder obstruction (Renal and urinary disorders) | 3 | 3
Bone marrow myelogram abnormal (Investigations) | 0 | 1
Bronchitis (Infections and infestations) | 3 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Cellulitis (Infections and infestations) | 3 | 9
Colitis (Gastrointestinal disorders) | 0 | 4
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Cystitis (Infections and infestations) | 1 | 1
Death (General disorders) | 2 | 3
Diverticular perforation (Gastrointestinal disorders) | 1 | 0
Face oedema (General disorders) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 | 1
Haemoglobin decreased (Investigations) | 3 | 9
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 3
IIIrd nerve disorder (Nervous system disorders) | 1 | 0
Influenza like illness (General disorders) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Maculopathy (Eye disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 2
Mouth ulceration (Gastrointestinal disorders) | 0 | 1
Mucosal inflammation (General disorders) | 1 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 7 | 13
Oedema (General disorders) | 0 | 1
Oesophageal infection (Infections and infestations) | 0 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 4 | 1
Peritonitis (Infections and infestations) | 1 | 1
Prostatic obstruction (Reproductive system and breast disorders) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 1
Sinus node dysfunction (Cardiac disorders) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 1
Tracheal obstruction (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 1
Anal fissure (Gastrointestinal disorders) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 2
Anastomotic leak (Injury, poisoning and procedural complications) | 0 | 1
Aphasia (Nervous system disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 7 | 4
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cellulitis of male external genital organ (Infections and infestations) | 0 | 1
Cerebral haematoma (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 3
Cerebrovascular accident (Nervous system disorders) | 4 | 2
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Dehydration (Metabolism and nutrition disorders) | 11 | 21
Depressed level of consciousness (Nervous system disorders) | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 5
Malaise (General disorders) | 0 | 1
Megacolon (Gastrointestinal disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neutrophil count (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 2 | 0
Oedema peripheral (General disorders) | 3 | 6
Peau d'orange (Skin and subcutaneous tissue disorders) | 0 | 1
Periodontal disease (Gastrointestinal disorders) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Renal impairment (Renal and urinary disorders) | 3 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 7
Subileus (Gastrointestinal disorders) | 1 | 0
Sudden death (General disorders) | 3 | 0
Transaminases increased (Investigations) | 1 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 | 3
Weight decreased (Investigations) | 1 | 1
Agranulocytosis (Blood and lymphatic system disorders) | 1 | 0
Ataxia (Nervous system disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 2 | 0
Cardiac arrest (Cardiac disorders) | 1 | 2
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 2 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Coma (Nervous system disorders) | 0 | 1
Disorientation (Psychiatric disorders) | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Endocarditis (Infections and infestations) | 0 | 1
Fatigue (General disorders) | 9 | 15
Femur fracture (Injury, poisoning and procedural complications) | 2 | 2
Gastric ulcer (Gastrointestinal disorders) | 3 | 2
Haematoma (Vascular disorders) | 0 | 1
Haemoglobin (Investigations) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 2
Infection (Infections and infestations) | 4 | 8
Lobar pneumonia (Infections and infestations) | 1 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Lung infection (Infections and infestations) | 0 | 2
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Monoplegia (Nervous system disorders) | 1 | 0
Multi-organ failure (General disorders) | 1 | 3
Nephrotic syndrome (Renal and urinary disorders) | 0 | 2
Neuralgia (Nervous system disorders) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 18 | 19
Oral candidiasis (Infections and infestations) | 1 | 1
Penile pain (Reproductive system and breast disorders) | 1 | 0
Performance status decreased (General disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 19
Proctalgia (Gastrointestinal disorders) | 0 | 1
Proctitis (Gastrointestinal disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 4
Sepsis (Infections and infestations) | 6 | 7
Tachycardia (Cardiac disorders) | 1 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Ureteric obstruction (Renal and urinary disorders) | 1 | 1
Ureteric stenosis (Renal and urinary disorders) | 0 | 1
Urinary bladder polyp (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 9 | 9
Urinary tract infection (Infections and infestations) | 7 | 10
Urinary tract obstruction (Renal and urinary disorders) | 2 | 3
Volvulus (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 6
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 3
Alanine aminotransferase increased (Investigations) | 0 | 1
Aortic dissection (Vascular disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder outlet obstruction (Renal and urinary disorders) | 0 | 1
Candida infection (Infections and infestations) | 0 | 1
Cardiac failure (Cardiac disorders) | 3 | 1
Central nervous system haemorrhage (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Clostridium test positive (Investigations) | 0 | 1
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 0 | 3
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
Gangrene (Infections and infestations) | 0 | 1
General physical health deterioration (General disorders) | 1 | 4
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 18 | 10
Haemorrhage (Vascular disorders) | 1 | 1
Herpes zoster (Infections and infestations) | 2 | 0
Hydrocele (Congenital, familial and genetic disorders) | 1 | 0
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Intestinal sepsis (Infections and infestations) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 2
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Motor dysfunction (Nervous system disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 2 | 2
Neutropenic sepsis (Infections and infestations) | 0 | 2
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 3
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 2
Peptic ulcer (Gastrointestinal disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 2
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0
Vasculitis (Vascular disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Amaurosis fugax (Eye disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 8 | 8
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Balanoposthitis infective (Infections and infestations) | 0 | 1
Chest pain (General disorders) | 8 | 9
Condition aggravated (General disorders) | 1 | 0
Depression suicidal (Psychiatric disorders) | 0 | 1
Device related infection (Infections and infestations) | 0 | 1
Embolism (Vascular disorders) | 1 | 0
Encephalitis (Infections and infestations) | 1 | 0
Enterocolitis bacterial (Infections and infestations) | 0 | 1
Fungal oesophagitis (Infections and infestations) | 1 | 0
Generalised oedema (General disorders) | 1 | 1
Haematemesis (Gastrointestinal disorders) | 2 | 0
Hepatic pain (Hepatobiliary disorders) | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 3
Ileus (Gastrointestinal disorders) | 1 | 0
Infarction (Vascular disorders) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Platelet count decreased (Investigations) | 1 | 0
Pneumonia (Infections and infestations) | 22 | 33
Procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 17 | 5
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 5 | 8
Renal failure (Renal and urinary disorders) | 5 | 5
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Septic shock (Infections and infestations) | 3 | 10
Supraventricular tachyarrhythmia (Cardiac disorders) | 0 | 1
Syncope (Nervous system disorders) | 5 | 4
Thrombosis (Vascular disorders) | 0 | 2
Urine output decreased (Investigations) | 0 | 1
Urosepsis (Infections and infestations) | 4 | 1
Vena cava thrombosis (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 1
Abscess intestinal (Infections and infestations) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 7
Bacteraemia (Infections and infestations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 2
Bronchopneumonia (Infections and infestations) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 3 | 1
Colorectal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 3
Diarrhoea (Gastrointestinal disorders) | 10 | 44
Disease progression (General disorders) | 0 | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 1
Gastrointestinal infection (Infections and infestations) | 1 | 3
Hypertension (Vascular disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 2 | 1
Intracranial pressure increased (Nervous system disorders) | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 1 | 0
Localised oedema (General disorders) | 1 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 3
Myocardial infarction (Cardiac disorders) | 1 | 2
Oedema genital (Reproductive system and breast disorders) | 1 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 2 | 0
Pneumonia streptococcal (Infections and infestations) | 0 | 1
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 9
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary venous thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 2
Testicular mass (Reproductive system and breast disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 10 | 14
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Anal abscess (Infections and infestations) | 2 | 1
Angina pectoris (Cardiac disorders) | 1 | 2
Anxiety (Psychiatric disorders) | 1 | 0
Appendicitis (Infections and infestations) | 3 | 1
Arrhythmia (Cardiac disorders) | 0 | 2
Asthenia (General disorders) | 7 | 13
Cardiac disorder (Cardiac disorders) | 0 | 1
Chills (General disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1
Confusional state (Psychiatric disorders) | 2 | 6
Constipation (Gastrointestinal disorders) | 10 | 5
Device related sepsis (Infections and infestations) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 1
Erysipelas (Infections and infestations) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 27 | 32
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 7 | 8
Gastrointestinal ulcer (Gastrointestinal disorders) | 1 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 6 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Neutropenic infection (Infections and infestations) | 3 | 3
Obstructive uropathy (Renal and urinary disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 6 | 11
Perirectal abscess (Infections and infestations) | 2 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 6 | 4
Spinal fracture (Injury, poisoning and procedural complications) | 3 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 3
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Urogenital haemorrhage (Renal and urinary disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=757) | Dasatinib (N=761)
Dyspepsia (Gastrointestinal disorders) | 59 | 50
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 127 | 154
Lacrimation increased (Eye disorders) | 86 | 48
Muscle spasms (Musculoskeletal and connective tissue disorders) | 42 | 15
Nail disorder (Skin and subcutaneous tissue disorders) | 119 | 80
Pain (General disorders) | 62 | 47
Pyrexia (General disorders) | 71 | 132
Stomatitis (Gastrointestinal disorders) | 47 | 47
Anaemia (Blood and lymphatic system disorders) | 142 | 217
Haemoglobin decreased (Investigations) | 27 | 49
Mucosal inflammation (General disorders) | 52 | 70
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 55 | 62
Nausea (Gastrointestinal disorders) | 231 | 288
Oedema (General disorders) | 47 | 36
Bone pain (Musculoskeletal and connective tissue disorders) | 70 | 61
Cough (Respiratory, thoracic and mediastinal disorders) | 112 | 137
Dehydration (Metabolism and nutrition disorders) | 23 | 44
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 41 | 33
Headache (Nervous system disorders) | 65 | 82
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 40 | 35
Oedema peripheral (General disorders) | 207 | 162
Weight decreased (Investigations) | 77 | 121
Fatigue (General disorders) | 329 | 334
Neutropenia (Blood and lymphatic system disorders) | 67 | 79
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 28 | 117
Rash (Skin and subcutaneous tissue disorders) | 75 | 106
Urinary tract infection (Infections and infestations) | 67 | 73
Abdominal pain (Gastrointestinal disorders) | 67 | 66
Dysgeusia (Nervous system disorders) | 147 | 165
Haematuria (Renal and urinary disorders) | 44 | 46
Pain in extremity (Musculoskeletal and connective tissue disorders) | 128 | 115
Alopecia (Skin and subcutaneous tissue disorders) | 326 | 311
Chest pain (General disorders) | 34 | 49
Insomnia (Psychiatric disorders) | 95 | 76
Myalgia (Musculoskeletal and connective tissue disorders) | 54 | 50
Neuropathy peripheral (Nervous system disorders) | 109 | 83
Peripheral sensory neuropathy (Nervous system disorders) | 106 | 98
Arthralgia (Musculoskeletal and connective tissue disorders) | 124 | 104
Back pain (Musculoskeletal and connective tissue disorders) | 194 | 148
Decreased appetite (Metabolism and nutrition disorders) | 151 | 207
Diarrhoea (Gastrointestinal disorders) | 312 | 414
Hypertension (Vascular disorders) | 42 | 22
Muscular weakness (Musculoskeletal and connective tissue disorders) | 51 | 38
Vomiting (Gastrointestinal disorders) | 117 | 166
Weight increased (Investigations) | 64 | 36
Asthenia (General disorders) | 143 | 163
Constipation (Gastrointestinal disorders) | 189 | 157
Dizziness (Nervous system disorders) | 61 | 64
Dry skin (Skin and subcutaneous tissue disorders) | 46 | 54
Hyperglycaemia (Metabolism and nutrition disorders) | 55 | 41
Hypocalcaemia (Metabolism and nutrition disorders) | 24 | 40
Paraesthesia (Nervous system disorders) | 59 | 44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.